CLINICAL TRIAL: NCT04874688
Title: Child Health, Agriculture and Integrated Nutrition (CHAIN): a Randomized Trial to Close the Nutrient Gap in Rural Zimbabwe
Brief Title: Child Health, Agriculture and Integrated Nutrition
Acronym: CHAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: CIMMYT (Unknown); University of Southampton (Other); Ministry of Health and Child Welfare, Zimbabwe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRCZ/A/2679
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Stunting
Keywords: Infant and young child feeding; Nutrients; Environmental enteric dysfunction; Microbiota; Immune function; Systemic inflammation; Metabolic profile
MeSH Terms: conditions — Growth Disorders | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Intervention Model Description: Individually randomized, unblinded clinical trial
Who Masked: Investigator
Masking Description: Families and fieldworkers measuring outcome measures are not blinded. Analysts and laboratory scientists will be blinded to intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IYCF-Only (Active Comparator): Infants in the IYCF-only arm will receive white maize and SQ-LNS daily from 6 months of age, and the primary caregiver will receive a series of behaviour-change modules delivered by village health workers.
  Interventions: Dietary Supplement: Small-quantity lipid-based nutrient supplement; Dietary Supplement: White maize meal
- IYCF-Plus (Experimental): Infants in the IYCF-plus arm will receive orange provitamin A-fortified maize and SQ-LNS daily from 6 months of age, plus powdered NUA-45 sugar beans, moringa leaf powder, and powdered whole egg; and the primary caregiver will receive a series of behaviour-change modules delivered by village health workers.
  Interventions: Dietary Supplement: Small-quantity lipid-based nutrient supplement; Dietary Supplement: Provitamin A biofortified maize; Dietary Supplement: NUA-45 biofortified sugar beans; Dietary Supplement: Moringa oleifera; Dietary Supplement: Whole egg powder

INTERVENTIONS:
Dietary Supplement: Small-quantity lipid-based nutrient supplement — Small Quantity Lipid-based Nutrient Supplement (SQ-LNS) is a food supplement rich in both macro and micronutrients (calories, proteins, fat and multivitamin mix). SQ-LNS is not considered a regulated drug product in Zimbabwe, or by the United States Food and Drug Administration (FDA). It is commercially available for prevention of chronic malnutrition, produced by Nutriset (https://www.nutriset.fr/products/en/enov-nutributter2). Each child will receive a daily sachet of 20g SQ-LNS between 6-12 months of age, consumed directly from the sachet or mixed with porridge.
Dietary Supplement: Provitamin A biofortified maize — Provitamin A Maize Meal is orange maize-meal processed from provitamin A-rich orange maize. PVA maize meal will be sourced from International Maize and Wheat Improvement Centre (CIMMYT). Children in the intervention arm will consume 13g - 128g of pro-vitamin A (PVA) maize meal, with added powders. Each family will receive a monthly ration of 5kg PVA maize and this ration takes into consideration of household sharing. Families with children in the IYCF arm will receive white maize meal.
  Other Names: Orange maize
  Arms: IYCF-Plus
Dietary Supplement: NUA-45 biofortified sugar beans — NUA 45 bean powder is ground from roasted iron and zinc-rich biofortified sugar beans. NUA 45 bean powder will be sourced from Sky Brands Ltd Company. Children will consume a daily dose of 5g - 15g of NUA 45 bean powder added to complementary foods.
  Arms: IYCF-Plus
Dietary Supplement: Moringa oleifera — Moringa oleifera is an edible plant abundant in dry tropic regions including Zimbabwe. It is known to be rich in micronutrients and has been widely used in Zimbabwe and around the world both as a food and a herb. Moringa oleifera leaf powder, is a dried and ground powder produced from Moringa oleifera leaves using traditional methods. It has been widely used to fortify complementary foods in the African region with the aim of improving micronutrient status. Moringa oleifera leaf powder will be sourced from Lemex Products Company. Children will receive a daily dose of 5g - 15g of Moringa leaf powder added to complementary foods.
  Other Names: Moringa leaf powder
  Arms: IYCF-Plus
Dietary Supplement: Whole egg powder — Egg Powder is hydrolysed non-genetically modified organism (GMO), fine and unflavoured whole egg powder. It is processed with no additives, preservatives, lecithin, added sugar, soy or monosodium glutamate. Egg powder will be sourced from France (A & D Food Ingredients - distributor in South Africa). Children in the IYCF-plus arm will receive a daily dose of 14g egg powder. A 15% extra amount of egg powder will be provided to families taking into consideration of household sharing. Egg powder will be provided in sealed plastic jars similar to that of peanut butter and households will receive promotion messages to store the powder in a cool, dry place and avoiding contact with water or moisture during use.
  Arms: IYCF-Plus
Dietary Supplement: White maize meal — Commercial white maize meal will be provided monthly. Infants age 6-8 months will receive 45g (3 tablespoons) daily; infants aged 9-12 months will receive 71g (4.5 tablespoons) daily.
  Arms: IYCF-Only

SUMMARY:
CHAIN is an open-label, individually randomized trial of improved infant and young child feeding (IYCF) versus "IYCF-plus" among 192 infants enrolled between 5-6 months of age in Shurugwi district, rural Zimbabwe. Interventions comprise sequential behaviour-change interventions delivered by village health workers together with food supplements. In the IYCF arm, infants will receive white maize and small-quantity lipid-based nutrient supplement (SQ-LNS) daily from 6 months of age. In the IYCF-plus arm, infants will receive orange pro-vitamin A-biofortified maize, and SQ-LNS, plus powdered sugar beans, moringa and whole egg powder. The primary outcome will be the proportion of infants in each trial arm reaching daily energy requirements at 9 months of age (visit window 9-11 months of age). Secondary outcomes are other nutrient intake, anthropometry and haemoglobin. Tertiary outcomes are laboratory measures of microbiome composition, environmental enteric dysfunction, inflammation, innate immune function, circulating choline and essential amino acids, and urinary metabolic profile. Two qualitative substudies will explore i) the feasibility and acceptability of the IYCF-plus intervention; and ii) the influence of migration on household food consumption and production.

DETAILED DESCRIPTION:
Linear growth failure (stunting) in childhood is the most prevalent form of undernutrition globally. Diets in rural sub-Saharan Africa have low dietary diversity and a reliance on white maize, which is high in starch and low in other nutrients. Improving infant and young child feeding (IYCF) during the period of complementary feeding from 6-24 months of age, including use of daily small-quantity lipid-based nutrient supplements (SQ-LNS), has a modest impact on linear growth. However, despite intensive IYCF interventions, infants often still have nutrient gaps. Furthermore, three key biological barriers (environmental enteric dysfunction, dysbiosis of the gut microbiota, and systemic inflammation) limit nutrient uptake and utilisation.

The overarching goal of this trial is to fill key nutrient gaps among infants in rural sub-Saharan Africa through an improved IYCF intervention using locally available foods that can ultimately be self-sustaining through agriculture. Addressing intake, uptake and utilization of nutrients in tandem, through use of 'functional foods' could ultimately improve growth and development in young children.

CHAIN is an open-label, individually randomized trial of improved infant and young child feeding (IYCF) versus "IYCF-plus" among 192 infants enrolled between 5-6 months of age in Shurugwi district, rural Zimbabwe. Interventions comprise sequential behaviour-change interventions delivered by village health workers together with food supplements. In the IYCF arm, infants will receive white maize and small-quantity lipid-based nutrient supplement (SQ-LNS) daily from 6 months of age. In the IYCF-plus arm, infants will receive orange pro-vitamin A-biofortified maize, and daily SQ-LNS, plus additional foods that are nutrient-rich, culturally acceptable and locally sustainable: NUA-45 biofortified sugar beans, moringa leaf powder and whole egg powder. For the duration of the trial, these foods will be provided as dried powders, which can be added to infant porridge as point-of-use fortificants. Together, these food supplements have the added plausible benefit of improving the microbiota and gut barrier function and reducing intestinal and systemic inflammation.

The primary outcome will be the proportion of infants in each trial arm reaching daily energy requirements at 9 months of age (visit window 9-11 months of age). Secondary outcomes are intake of protein, iron, zinc and folate; height-for-age Z score, weight-for-age Z-score, and weight-for-height Z-score; and haemoglobin. Tertiary outcomes are laboratory measures of microbiome composition, environmental enteric dysfunction, inflammation, innate immune function, circulating choline and essential amino acids, and urinary metabolic profile. Two qualitative substudies will explore i) the feasibility and acceptability of the IYCF-plus intervention; and ii) the influence of migration on household food consumption and production.

Trained research nurses will collect baseline data on maternal and infant demographics, nutritional status and household characteristics. Infants will have anthropometry measurements undertaken, and baseline infant stool, urine and blood samples will be collected by the research nurse.

All interventions are delivered by trained village health workers, each of whom has an allocated catchment area as part of their regular duties. VHW will provide regular interactive education modules for the IYCF and IYCF-plus arms, and deliver monthly supplies of food supplements from enrolment until 12 months of infant age. VHW will be overseen by a cadre of intervention nurses, who will provide supportive supervision, conduct spot checks, and hold meetings with the VHWs they supervise to ensure consistency in delivering the trial messages. In this way, the cadre delivering the interventions (VHW, supervised by intervention nurses) will be separated from the cadre measuring the trial outcomes (research nurses), to avoid courtesy bias among participants.

At the endline home visit at 9 months of infant age (window: 9-11 months) a research nurse will collect data by maternal recall on use of the IYCF or IYCF-plus supplements and on infant dietary intake by multi-pass 24-hour dietary recall. Infants will have repeat anthropometry undertaken, and urine, stool and blood samples collected, with point-of-care measurement of haemoglobin. A further visit will be undertaken 1 week later in 50% of households to repeat the 24-hour diet recall.

Laboratory analyses will include measures of environmental enteric dysfunction; microbiome composition; innate immune function; systemic inflammation; circulating choline and essential amino acids; and urinary metabolic profile.

To explore the feasibility and acceptability of the IYCF-plus intervention, one qualitative substudy will collect information from study households, the village health workers who support them, and key community stakeholders. Research findings will inform how this intervention can be rolled out at scale. Up to 20 households will be purposively sampled after the baseline survey. In-depth interviews will be conducted by a trained social scientist when the infant is 7-9 months old after the households have been introduced to all the nutrients (SQ-LNS and food powders), focused on household feeding practices and norms, household farming practices and related livelihood strategies, and the acceptability of the new supplements. Attention will also be focused on the influence of gendered norms and social relations on household decision-making practices in these areas.

To identify the influence of migration on household food consumption and production, a second qualitative substudy will enrol up to 30 participating households identified from the baseline questionnaire survey as having at least one family member who has migrated. In addition to exploring the impact of migration on household food consumption and production practices, the in-depth interviews conducted for this sub-study aim to investigate possible interactions between migration and household participation in the CHAIN intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5-6 months
* Planning to live in the study area for the duration of the trial

Exclusion Criteria:

* Severe infant disability that interferes with feeding
* Known allergy to peanuts or eggs

Ages: 5 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Energy intake | 9 months of age (window 9-11 months)
  Percentage of infants meeting daily energy requirements, measured by multi-pass 24-hour dietary recall,

SECONDARY OUTCOMES:
Protein intake | 9 months of age (window 9-11 months)
  Percentage of infants meeting daily protein requirements at 9 months of age, measured by multi-pass 24-hour dietary recall
Iron intake | 9 months of age (window 9-11 months)
  Percentage of infants meeting daily iron requirements at 9 months of age, measured by multi-pass 24-hour dietary recall
Zinc intake | 9 months of age (window 9-11 months)
  Percentage of infants meeting daily zinc requirements at 9 months of age, measured by multi-pass 24-hour dietary recall
Folate intake | 9 months of age (window 9-11 months)
  Percentage of infants meeting daily folate requirements at 9 months of age, measured by multi-pass 24-hour dietary recall
Height-for-age Z-score | 9 months of age (window 9-11 months)
  Height-for-age expressed as a Z-score compared to the World Health Organization 2006 reference median
Weight-for-age Z score | 9 months of age (window 9-11 months)
  Weight-for-age expressed as a Z-score compared to the World Health Organization 2006 reference median
Weight-for-height Z score | 9 months of age (window 9-11 months)
  Weight-for-height expressed as a Z-score compared to the World Health Organization 2006 reference median
Haemoglobin | 9 months of age (window 9-11 months)
  Concentration of haemoglobin (in g/dL) in a whole blood finger prick sample, measured by HemoCue point-of-care assay and adjusted for altitude

OTHER OUTCOMES:
Microbiome maturity | 9 months of age (window 9-11 months)
  Microbiota-for-age Z-score
Environmental enteric dysfunction | 9 months of age (window 9-11 months)
  Biomarkers of intestinal inflammation (faecal neopterin and myeloperoxidase), small intestinal damage (plasma intestinal fatty acid binding protein, and citrulline), intestinal permeability (faecal alpha-1 antitrypsin), microbial translocation (plasma soluble CD14, lipopolysaccharide binding protein), systemic inflammation (plasma C-reactive protein, Alpha-1 acid hlycoprotein, tumour necrosis factor alpha and kynurenine-tryptophan ratio) and growth hormone axis (insulin-like growth factor 1), which will be analysed individually and then analysed in combination using principal components analysis to reduce data.
Innate immune cell phenotype | 9 months of age (window 9-11 months)
  Surface marker expression by peripheral blood monocytes and neutrophils
Innate immune cell function | 9 months of age (window 9-11 months)
  Surface marker expression and cytokine secretion from innate immune cells challenged with lipopolysaccharide in vitro relative to unstimulated controls
  Capacity of innate immune cells to internalise bacteria in vitro
Plasma essential amino acids | 9 months of age (window 9-11 months)
  Plasma concentrations of phenylalanine, valine, threonine, tryptophan, methionine, leucine, isoleucine, lysine and histidine, as measured by LC-MS-MS
Plasma choline | 9 months of age (window 9-11 months)
  Plasma concentration of choline, as measured by liquid chromatography with tandem mass spectrometry (LC-MS-MS)
Urinary metabolic signature | 9 months of age (window 9-11 months)
  Global untargeted metabolomic phenotyping undertaken by proton nuclear magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Smith, PhD, Principal Investigator — Zvitambo Institute for Maternal and Child Health Research
Locations (1):
- Zvitambo Institute for Maternal and Child Health Research, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available for sharing upon review of a request to the investigator team
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after primary analysis is completed

REFERENCES:
- [Derived] Smith LE, Chagwena DT, Bourke C, Robertson R, Fernando S, Tavengwa NV, Cairns J, Ndhlela T, Matumbu E, Brown T, Datta K, Mutasa B, Tengende A, Chidhanguro D, Langhaug L, Makanza M, Chasekwa B, Mutasa K, Swann J, Kelly P, Ntozini R, Prendergast A. Child Health, Agriculture and Integrated Nutrition (CHAIN): protocol for a randomised controlled trial of improved infant and young child feeding in rural Zimbabwe. BMJ Open. 2022 Dec 30;12(12):e056435. doi: 10.1136/bmjopen-2021-056435. PMID 36585147
- See also: Study protocol, intervention materials, statistical analysis plan and CRFs will be posted on this Open Science Framework site — https://osf.io/njy2a/